CLINICAL TRIAL: NCT04573322
Title: Open-label, Pharmacokinetic, Pharmacodynamic, Ascending Dose Safety lead-in Followed by a Single-center, Placebo-controlled, Double-blind, Adaptive, Safety and Efficacy, Pilot Study of Trans Sodium Crocetinate (TSC) in SARS-CoV-2 Infected Subjects
Brief Title: Safety and Efficacy of Trans Sodium Crocetinate (TSC) in SARS-CoV-2 (COVID-19) Infected Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Diffusion Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100-303
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Results first posted 2022-04-01 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: SARS-CoV-2 (Covid19)
Keywords: Hypoxemia; Hypoxia
MeSH Terms: conditions — COVID-19; Hypoxia | interventions — trans-sodium crocetinate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Open-label, pharmacokinetic, pharmacodynamic, ascending dose, safety and tolerability lead-in Single-center, randomized, placebo-controlled, double-blind, adaptive, safety and efficacy pilot
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Lead-in: no masking. Randomized pilot: The participants, care providers, investigators, and outcomes assessors are masked. The pharmacist, unblinded clinical research associate, and unblinded study drug administrator are not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Lead-in 0.25 mg/kg (Experimental): 0.25 mg/kg TSC, administered via IV bolus every 6 hours for up to 15 days
  Interventions: Drug: Trans Sodium Crocetinate
- Lead-in 0.50 mg/kg (Experimental): 0.50 mg/kg TSC, administered via IV bolus every 6 hours for up to 15 days
  Interventions: Drug: Trans Sodium Crocetinate
- Lead-in 1.0 mg/kg (Experimental): 1.0 mg/kg TSC, administered via IV bolus every 6 hours for up to 15 days
  Interventions: Drug: Trans Sodium Crocetinate
- Lead-in 1.5 mg/kg (Experimental): 1.5 mg/kg TSC, administered via IV bolus every 6 hours for up to 15 days
  Interventions: Drug: Trans Sodium Crocetinate
- Randomized Active TSC (Experimental): TSC, at the optimum safe and tolerable dose determined in the lead-in phase, administered via IV bolus every 6 hours for up to 15 days
  Interventions: Drug: Trans Sodium Crocetinate
- Randomized Placebo (Placebo Comparator): Normal Saline, in an equivalent volume by participant body weight, administered via IV bolus every 6 hours for up to 15 days
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Trans Sodium Crocetinate — TSC, at the optimum safe and tolerable dose determined in the lead-in phase, administered via IV bolus every 6 hours for up to 15 days
  Other Names: TSC
  Arms: Lead-in 0.25 mg/kg; Lead-in 0.50 mg/kg; Lead-in 1.0 mg/kg; Lead-in 1.5 mg/kg; Randomized Active TSC
Drug: Normal saline — Normal Saline, in an equivalent volume by participant body weight, administered via IV bolus every 6 hours for up to 15 days
  Other Names: 0.9% Sodium Chloride (NaCl)
  Arms: Randomized Placebo

SUMMARY:
This study will assess the safety and efficacy of TSC as a treatment for participants who are infected with SARS-CoV-2 (COVID-19).

DETAILED DESCRIPTION:
This trial has two phases. The first phase is an open-label, pharmacokinetic, pharmacodynamic, ascending dose, safety and tolerability lead-in. The second phase is a single-center, randomized, placebo-controlled, double-blind, adaptive, safety and efficacy, pilot.

The lead-in phase will study 4 doses of TSC and enroll 24 participants. Each TSC dose will be administered as an IV bolus injection to 6 unique participants per dose level administered four times per day (every 6 hours) for 5 days. Participants will be assigned in groups of 3, and a Safety Monitoring Committee (SMC) will review Dose Limiting Toxicities (DLTs) after each group of 3 participants. The first group of 3 participants will receive TSC at a dose of 0.25 mg/kg. If there are no DLTs, 3 additional subjects will be studied at 0.25 mg/kg. If there are 0 or 1 DLT among the 6 participants studied at 0.25mg/kg, 3 additional participants will be studied at the next higher dose, 0.5 mg/kg. If there are no DLTs an additional 3 participants will be studied at 0.5 mg/kg. If there are 0 or 1 DLTs among the 6 subjects studied at 0.5 mg/kg, 3 additional participants will be studied at the next higher dose, 1.0 mg/kg. The study will continue in this fashion seeking an observed toxicity rate that is < 0.33 among 6 participants at any one dose level, or TSC at 1.5 mg/kg proves to be safe and tolerable.

As participants complete the initial 5 days of treatment they will continue at their assigned TSC dose four times per day (every 6 hours) for up to 15 days. Participants will be assigned to dose levels in ascending order. The dose range is as follows.

* 0.25 mg/kg TSC + Standard of Care
* 0.50 mg/kg TSC + Standard of Care
* 1.00 mg/kg TSC + Standard of Care
* 1.50 mg/kg TSC + Standard of Care

At the completion of the lead-in the Safety Monitoring Committee (SMC) will examine the resultant safety and blood oxygenation (S:F) data for all participants and determine the optimum, safe and tolerable dose of TSC for use in the pilot study.

Dose Limiting Toxicity (DLT) is defined as any study drug related grade 3 or 4 adverse event during the treatment period, with the exception of pulmonary events in the CTCAE that are known complications of SARS-CoV-2 infection: Acute Respiratory Distress Syndrome (ARDS), Cough, Dyspnea, Hypoxia, Pneumonitis, Pulmonary Edema, Respiratory Failure, or Respiratory, Thoracic and Mediastinal disorders - Other. The SMC will apply clinical judgement in their review of adverse events (particularly abnormal laboratory results).

The two arm, randomized pilot will enroll up to 200 participants, and will be overseen by a Data Safety Monitoring Board (DSMB). TSC dosing will be at the selected optimum, safe and tolerable biologic dose with an active to placebo ratio of 2:1 toward providing the maximum potential benefit to participants. If two doses of TSC are to be studied in the randomized pilot the active to placebo ratio will be 2:2:1. Randomization will be stratified by disease severity, age and presence of pre-specified comorbidities. The treatment arms are as follows.

* TSC + Standard of Care
* Placebo + Standard of Care

Each TSC dose will be administered as an IV bolus injection 4 times per day (every 6 hours) for up to 15 days. Participants randomized to placebo will receive an IV bolus injection of an equivalent volume by participant weight of Normal Saline four times per day (every 6 hours) for up to 15 days.

All study drug administration will be performed by unblinded medical staff. Participants, investigators and caregivers will not see the injection or injection site or be aware of randomization.

Blood oxygenation will be measured via recorded continuous pulse oximetry and the SpO2:Fraction of Inspired Oxygen (FiO2) ratio calculated.

All participants will undergo safety and efficacy assessments including laboratory assays, blood sampling on days 1 through day 15 (while hospitalized) and day 29 by return clinic visit or if still hospitalized.

All participants, whether a part of the lead-in phase or randomized pilot, will be assessed for survival, serious adverse events and adverse events by requested return to the clinic on Day 60.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized subjects with confirmed SARS-CoV-2 infection and hypoxemia, defined as SpO2 < 94% on room air or requiring supplemental oxygen
2. Laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen < 72 hours prior to enrollment.
3. WHO ordinal scale score of 3, 4 or 5 at baseline
4. Male or non-pregnant female adult ≥18 years of age at time of enrolment.
5. Subject (or legally authorized representative (LAR)) provides written informed consent prior to initiation of any study procedures.
6. Understands and agrees to comply with planned study procedures.
7. Illness of any duration
8. Women of childbearing potential must have a negative blood pregnancy test at the screening/baseline visit (Day 1) and agree to use a double method of birth control through 30 days after the last dose of study drug.

Exclusion Criteria:

1. Intubated and mechanically ventilated at baseline
2. Receiving extracorporeal membrane oxygenation (ECMO) at baseline
3. Severe organ dysfunction (SOFA score > 10)
4. Patient or LAR unable to provide written informed consent
5. ALT/AST > 3 times the upper limit of normal or serum bilirubin > 1.5 times the upper limit of normal
6. Estimated glomerular filtration rate (eGFR) by Modification of Diet in Renal Disease (MDRD) formula < 30 mL/min/1.73 m^2 or on dialysis
7. Pregnancy or breast feeding.
8. Anticipated transfer to another hospital which is not a study site within 72 hours.
9. Allergy to any study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Streinu Cercel, MD, Principal Investigator — National Institute of Infectious Diseases, Bucharest, Romania
Locations (1):
- National Institute of Infectious Diseases- Prof. Dr. Matei Balş, Bucharest, Romania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1 lead-in was conducted; however, the study was completed prior to initiation of Phase 2. Therefore, only data are reported for the lead-in phase, as no data were collected for Phase 2.
Period: Overall Study
Arm/Group | Lead-in 0.25 mg/kg | Lead-in 0.50 mg/kg | Lead-in 1.0 mg/kg | Lead-in 1.5 mg/kg
Started | 6 | 6 | 7 | 6
Completed | 5 | 4 | 5 | 3
Not Completed | 1 | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Phase 1 lead-in was conducted; however, the study was completed prior to initiation of Phase 2. Therefore, only data are reported for the lead-in phase, as no data were collected for Phase 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lead-in 0.25 mg/kg | Lead-in 0.50 mg/kg | Lead-in 1.0 mg/kg | Lead-in 1.5 mg/kg | Total
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7 | 5 | 19
  >=65 years | 2 | 3 | 0 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.50 (18.87) | 60.83 (16.04) | 54.43 (8.16) | 57.50 (8.89) | 56.00 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 4 | 13
  Male | 3 | 4 | 3 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 7 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 6 | 6 | 7 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: Lead-in phase: Overall summary of subjects with TEAEs
Time Frame: Up to 70 days post-study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in 0.25 mg/kg | Lead-in 0.50 mg/kg | Lead-in 1.0 mg/kg | Lead-in 1.5 mg/kg
Number analyzed (Participants) | 6 | 6 | 7 | 6
Participants
  Patients with any TEAE | 3 | 4 | 5 | 2
  Patients with any Serious TEAE | 1 | 1 | 0 | 0
  Patients with any TEAE of DLT | 0 | 0 | 0 | 0
  Patients with any TEAE Resulting in Death | 1 | 0 | 0 | 0
  Patients with any TEAE Leading to Study Drug Discontinuation | 0 | 1 | 0 | 0
  Patients with any TEAE Leading to Study Drug Interruption | 0 | 0 | 0 | 0
  Patients with any TEAE with CTCAE Grade 3 or 4 | 1 | 3 | 0 | 1

2. Primary Outcome: Time to Recovery Through Day 28
Description: Lead-in phase: Time to achieve (and maintain through Day 28) a World Health Organization (WHO) ordinal COVID-19 severity scale score of 1, 2 or 3 with a minimum 1-point improvement from baseline. The scale assesses clinical status and the range is 0-8, as follows:
  0. Uninfected - No clinical or virological evidence of infection
  1. Ambulatory - No limitation of activities
  2. Ambulatory - Limitation of activities
  3. Hospitalized, Mild Disease - Hospitalized, no oxygen therapy
  4. Hospitalized, Mild Disease - Oxygen by mask or nasal prongs
  5. Hospitalized Severe Disease - Non-invasive ventilation or high-low oxygen
  6. Hospitalized Severe Disease - Intubation and mechanical ventilation
  7. Hospitalized Severe Disease - Ventilation + additional organ support (pressors, Renal Replacement Therapy (RRT), Extracorporeal Membrane Oxygenation (ECMO)
  8. Dead - Death
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lead-in 0.25 mg/kg | Lead-in 0.50 mg/kg | Lead-in 1.0 mg/kg | Lead-in 1.5 mg/kg
Number analyzed (Participants) | 6 | 6 | 7 | 6
days | 14.33 (11.54) | 13.67 (8.43) | 7.71 (4.31) | 7.50 (1.22)

3. Secondary Outcome: Change From Baseline in WHO Ordinal Severity Scale as a Categorical Improvement or Worsening
Description: Lead-in phase: Number and percentage of patients by WHO Severity Scale change from baseline through Day 7
  World Health Organization (WHO) Ordinal Severity Scale
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, no requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow O2
  6. Hospitalized, on invasive mechanical ventilation or ECMO
  7. Death
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in 0.25 mg/kg | Lead-in 0.50 mg/kg | Lead-in 1.0 mg/kg | Lead-in 1.5 mg/kg
Number analyzed (Participants) | 6 | 6 | 7 | 6
Participants
  1 Point Worse from Day 1 to Day 7 | 0 | 1 | 0 | 0
  No Change from Day 1 to Day 7 | 3 | 3 | 5 | 1
  1 Point Improvement from Day 1 to Day 7 | 1 | 2 | 1 | 5
  No Data Collected on Day 7 | 2 | 0 | 1 | 0

4. Secondary Outcome: Oxygenation - Ventilator Free Days
Description: Lead-in phase: Ventilator free days in the first 28 days (to day 29).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lead-in 0.25 mg/kg | Lead-in 0.50 mg/kg | Lead-in 1.0 mg/kg | Lead-in 1.5 mg/kg
Number analyzed (Participants) | 6 | 6 | 7 | 6
days | 19.7 (6.05) | 16.00 (5.33) | 15.43 (7.28) | 19.83 (1.17)

5. Secondary Outcome: Hospital Length of Stay
Description: Lead-in phase: Days of treatment during the inpatient period
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lead-in 0.25 mg/kg | Lead-in 0.50 mg/kg | Lead-in 1.0 mg/kg | Lead-in 1.5 mg/kg
Number analyzed (Participants) | 6 | 6 | 7 | 6
days | 8.67 (2.66) | 9.67 (2.88) | 8.57 (3.78) | 8.00 (2.19)

6. Secondary Outcome: Oxygenation - Time to Return to Baseline
Description: Lead-in phase: Time to return to room air or baseline oxygen requirement
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lead-in 0.25 mg/kg | Lead-in 0.50 mg/kg | Lead-in 1.0 mg/kg | Lead-in 1.5 mg/kg
Number analyzed (Participants) | 6 | 6 | 7 | 6
days | 7.50 (5.68) | 18.92 (18.25) | 11.79 (7.47) | 5.50 (2.45)

7. Secondary Outcome: Oxygenation - Pulse Oximetry
Description: Lead-in phase: Blood oxygenation by recorded continuous pulse oximetry (SpO2:FiO2 ratio)
Time Frame: Baseline through Day 10
Population: There are some time points where data were not collected and, for the later timepoints, subjects discontinued.
Measure: Mean (Standard Deviation); unit: SpO2:FiO2
Arm/Group | Lead-in 0.25 mg/kg | Lead-in 0.50 mg/kg | Lead-in 1.0 mg/kg | Lead-in 1.5 mg/kg
Number analyzed (Participants) | 6 | 6 | 7 | 6
SpO2:FiO2
  Baseline (Pre First Dose) | 261.83 (73.80) | 164.33 (64.91) | 183.97 (41.34) | 255.03 (57.54)
  Day 1, Prior to Dose 1 | 261.83 (73.80) | 164.33 (64.91) | 183.97 (41.34) | 255.03 (57.54)
  Day 1, 1 Minute Post Dose 1 | 261.22 (74.87) | 163.33 (61.87) | 189.16 (46.07) | 255.33 (57.03)
  Day 1, 10 Minutes Post Dose 1 | 261.22 (74.90) | 164.87 (63.89) | 188.37 (46.00) | 255.15 (55.76)
  Day 1, 30 Minutes Post Dose 1 | 260.73 (76.50) | 165.67 (63.91) | 187.81 (45.89) | 256.07 (56.38)
  Day 1, 1.5 Hours Post Dose 1 | 263.22 (76.78) | 164.32 (62.38) | 187.89 (45.01) | 255.65 (54.28)
  Day 1, 3 Hours Post Dose 1 | 262.82 (78.20) | 165.20 (62.96) | 189.80 (46.50) | 256.67 (55.38)
  Day 1, Prior to Dose 2 | 252.98 (87.49) | 165.35 (63.48) | 188.84 (45.79) | 255.95 (56.01)
  Day 1, Prior to Dose 3 | 253.23 (89.57) | 166.17 (61.57) | 189.86 (43.19) | 255.72 (54.41)
  Day 1, Prior to Dose 4 | 252.47 (88.97) | 165.83 (64.40) | 189.40 (44.72) | 255.78 (55.36)
  Day 2, Prior to Dose 1 | 274.90 (118.47) | 165.32 (63.52) | 207.80 (30.76) | 275.20 (51.66)
  Day 2, 1 Minute Post Dose 1: number analyzed (Participants) | 6 | 6 | 3 | 0
  Day 2, 1 Minute Post Dose 1 | 270.90 (118.00) | 165.98 (63.00) | 202.00 (33.54) |
  Day 2, Prior to Dose 2: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 2, Prior to Dose 2 | 303.17 (147.94) | 172.12 (93.68) | 201.52 (39.10) | 267.90 (58.71)
  Day 2, Prior to Dose 3: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 2, Prior to Dose 3 | 300.43 (146.10) | 173.68 (94.74) | 204.42 (49.32) | 267.57 (56.69)
  Day 2, Prior to Dose 4: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 2, Prior to Dose 4 | 300.40 (147.32) | 174.33 (96.09) | 215.25 (39.84) | 266.48 (55.31)
  Day 3, Prior to Dose 1: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 3, Prior to Dose 1 | 265.12 (121.86) | 174.08 (95.67) | 247.23 (65.92) | 270.38 (71.65)
  Day 3, 1 Minute Post Dose 1: number analyzed (Participants) | 6 | 6 | 3 | 0
  Day 3, 1 Minute Post Dose 1 | 265.57 (121.88) | 174.08 (95.67) | 245.97 (71.98) |
  Day 3, Prior to Dose 2: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 3, Prior to Dose 2 | 265.47 (121.09) | 174.50 (93.34) | 248.12 (66.38) | 271.20 (71.78)
  Day 3, Prior to Dose 3: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 3, Prior to Dose 3 | 266.68 (120.38) | 175.05 (95.16) | 254.85 (60.32) | 271.70 (72.17)
  Day 3, Prior to Dose 4: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 3, Prior to Dose 4 | 260.48 (121.26) | 175.18 (95.25) | 259.87 (52.29) | 279.78 (67.28)
  Day 4, Prior to Dose 1: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 4, Prior to Dose 1 | 305.20 (147.31) | 179.77 (95.57) | 286.12 (95.93) | 321.28 (69.97)
  Day 4, Prior to Dose 2: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 4, Prior to Dose 2 | 304.03 (145.69) | 176.32 (87.93) | 264.70 (51.29) | 322.13 (71.91)
  Day 4, Prior to Dose 3: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 4, Prior to Dose 3 | 303.78 (144.73) | 176.32 (87.96) | 266.77 (53.24) | 320.35 (70.77)
  Day 4, Prior to Dose 4: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 4, Prior to Dose 4 | 303.85 (143.53) | 177.28 (89.45) | 302.93 (91.27) | 335.45 (59.25)
  Day 5, Prior to Dose 1: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 5, Prior to Dose 1 | 288.23 (151.89) | 176.55 (90.15) | 301.43 (91.31) | 343.87 (57.80)
  Day 5, Prior to Dose 2: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 5, Prior to Dose 2 | 288.03 (152.74) | 175.73 (88.43) | 316.25 (85.00) | 344.85 (56.57)
  Day 5, Prior to Dose 3: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 5, Prior to Dose 3 | 287.75 (151.69) | 176.88 (89.80) | 314.82 (82.17) | 355.35 (63.60)
  Day 5, Prior to Dose 4: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 5, Prior to Dose 4 | 288.23 (151.77) | 184.67 (102.13) | 297.18 (45.15) | 348.40 (75.66)
  Day 6, Prior to Dose 1: number analyzed (Participants) | 5 | 6 | 5 | 4
  Day 6, Prior to Dose 1 | 277.96 (175.22) | 189.23 (108.10) | 343.86 (68.07) | 341.25 (87.32)
  Day 6, Prior to Dose 2: number analyzed (Participants) | 2 | 4 | 5 | 4
  Day 6, Prior to Dose 2 | 303.55 (237.38) | 232.48 (138.43) | 322.44 (29.39) | 340.63 (90.97)
  Day 6, Prior to Dose 3: number analyzed (Participants) | 2 | 4 | 5 | 4
  Day 6, Prior to Dose 3 | 298.80 (230.66) | 233.93 (140.79) | 322.28 (27.37) | 356.63 (111.05)
  Day 6, Prior to Dose 4: number analyzed (Participants) | 2 | 4 | 5 | 4
  Day 6, Prior to Dose 4 | 301.90 (233.06) | 232.73 (138.10) | 343.38 (69.97) | 415.68 (95.68)
  Day 7, Prior to Dose 1: number analyzed (Participants) | 4 | 6 | 6 | 6
  Day 7, Prior to Dose 1 | 223.05 (99.73) | 236.05 (179.16) | 341.35 (67.98) | 433.48 (79.04)
  Day 7, Prior to Dose 2: number analyzed (Participants) | 2 | 3 | 4 | 3
  Day 7, Prior to Dose 2 | 218.85 (123.67) | 232.17 (212.20) | 371.78 (57.66) | 402.50 (115.29)
  Day 7, Prior to Dose 3: number analyzed (Participants) | 2 | 3 | 4 | 3
  Day 7, Prior to Dose 3 | 218.15 (124.66) | 223.37 (217.08) | 340.00 (11.55) | 403.43 (113.68)
  Day 7, Prior to Dose 4: number analyzed (Participants) | 2 | 3 | 4 | 3
  Day 7, Prior to Dose 4 | 219.60 (122.61) | 226.13 (214.31) | 401.85 (70.12) | 411.63 (91.25)
  Day 8, Prior to Dose 1: number analyzed (Participants) | 3 | 5 | 5 | 4
  Day 8, Prior to Dose 1 | 300.37 (164.58) | 187.60 (156.67) | 378.26 (85.71) | 425.80 (81.80)
  Day 8, Prior to Dose 2: number analyzed (Participants) | 2 | 3 | 3 | 1
  Day 8, Prior to Dose 2 | 220.30 (121.62) | 233.23 (206.81) | 422.60 (59.76) | 306.30
  Day 8, Prior to Dose 3: number analyzed (Participants) | 2 | 3 | 3 | 1
  Day 8, Prior to Dose 3 | 216.55 (122.40) | 248.03 (193.52) | 385.00 (75.75) | 306.30
  Day 8, Prior to Dose 4: number analyzed (Participants) | 2 | 3 | 2 | 1
  Day 8, Prior to Dose 4 | 219.70 (126.85) | 246.00 (191.24) | 410.15 (79.97) | 461.90
  Day 9, Prior to Dose 1: number analyzed (Participants) | 2 | 4 | 4 | 1
  Day 9, Prior to Dose 1 | 294.75 (229.60) | 221.45 (166.65) | 395.48 (79.54) | 461.90
  Day 9, Prior to Dose 2: number analyzed (Participants) | 2 | 3 | 2 | 1
  Day 9, Prior to Dose 2 | 291.25 (234.55) | 248.47 (189.04) | 398.35 (96.66) | 457.10
  Day 9, Prior to Dose 3: number analyzed (Participants) | 2 | 2 | 2 | 1
  Day 9, Prior to Dose 3 | 293.35 (231.58) | 149.95 (18.88) | 395.95 (93.27) | 457.10
  Day 9, Prior to Dose 4: number analyzed (Participants) | 2 | 2 | 2 | 1
  Day 9, Prior to Dose 4 | 291.70 (227.26) | 158.10 (28.43) | 471.40 (0.00) | 457.10
  Day 10, Prior to Dose 1: number analyzed (Participants) | 2 | 3 | 4 | 1
  Day 10, Prior to Dose 1 | 213.80 (130.81) | 154.67 (23.93) | 395.03 (82.81) | 457.10
  Day 10, Prior to Dose 2: number analyzed (Participants) | 2 | 2 | 2 | 1
  Day 10, Prior to Dose 2 | 214.50 (129.82) | 159.20 (31.96) | 394.30 (95.60) | 452.40
  Day 10, Prior to Dose 3: number analyzed (Participants) | 1 | 2 | 2 | 1
  Day 10, Prior to Dose 3 | 122.70 | 159.90 (30.97) | 469.05 (3.32) | 461.90
  Day 10, Prior to Dose 4: number analyzed (Participants) | 1 | 2 | 2 | 1
  Day 10, Prior to Dose 4 | 122.70 | 158.50 (32.95) | 469.05 (3.32) | 466.70

ADVERSE EVENTS:
Time Frame: AEs were collected for up to 70 days from the start of study drug administration through the 60-day follow-up visit (+10d).
Description: Phase 1 lead-in was conducted; however, the study was completed prior to initiation of Phase 2. Therefore, only data are reported for the lead-in phase, as no data were collected for Phase 2.
Arm/Group | Lead-in 0.25 mg/kg | Lead-in 0.50 mg/kg | Lead-in 1.0 mg/kg | Lead-in 1.5 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/6 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 4/6 | 5/7 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in 0.25 mg/kg (N=6) | Lead-in 0.50 mg/kg (N=6) | Lead-in 1.0 mg/kg (N=7) | Lead-in 1.5 mg/kg (N=6)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in 0.25 mg/kg (N=6) | Lead-in 0.50 mg/kg (N=6) | Lead-in 1.0 mg/kg (N=7) | Lead-in 1.5 mg/kg (N=6)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congestive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excessive Cerumen Production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernial Eventration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular Injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection Fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superinfection Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection Fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema Peripheral (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT04573322/Prot_SAP_000.pdf